CLINICAL TRIAL: NCT05023954
Title: mSEP: Investigation of Maternal Immunity and Testing of Physiological and Immune-metabolic Blood Markers for Maternal Sepsis
Brief Title: mSEP: Testing of Physiological and Immune-metabolic Blood Markers for Maternal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiff University (Other)
Collaborators: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: 262062version2
Record Dates: First submitted 2021-08-10; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Sepsis; Maternal Sepsis; Maternal Sepsis During Labor; SIRS; Pregnancy; Infection
MeSH Terms: conditions — Sepsis; Pregnancy Complications, Infectious | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: A longitudinal observational study looking at the pregnancy journey of 200 women Bloods taken for sepsis biomarkers including a genomic sepsis-test throughout the pregnancy journey
  Interventions: Diagnostic Test: Blood test
- B: A consecutive collection of data from 100 pregnant women with suspected sepsis Bloods taken for Sepsis Biomarkers including a genomic sepsis-test throughout the sepsis episode
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Drop of blood for RNA and metabolic analysis

SUMMARY:
A prospective observational cohort study investigating physiological parameters vs biological markers of whole blood in septic and non-septic pregnant woman to predict systemic immune health

DETAILED DESCRIPTION:
The altered physiology of pregnancy makes the signs and symptoms of sepsis less distinctive in the pregnant population. This can lead to both over treatment (with antibiotics) and late identification of sepsis. The progression of sepsis can be rapid in this population, resulting in severe morbidity and mortality. The mortality associated with sepsis in the general population is over 10%, while septic shock can increase this figure up to 30%. A study looking at maternal mortality due to sepsis recognised that the time from the onset of infection to death was less than 24 hours in 50% of patients. A review of the literature shows that half of the fatal cases of maternal sepsis could have been prevented with early detection of sepsis.

The unmet need is therefore a diagnostic bedside tool that can be performed on women identified as high risk via physiological parameters. The tool needs to be quick and easy to use whilst accurate at diagnosing sepsis.

Study Objectives

To evaluate the effectiveness of physiological parameters in predicting maternal sepsis.

To evaluate the effectiveness of alternative biomarkers in diagnosing maternal sepsis including a genomic sepsis-test.

Investigation of the systemic immune health of women undergoing an uncomplicated pregnancy and labour.

ELIGIBILITY:
Inclusion Criteria:

Pregnant with viable pregnancy confirmed on ultrasound at dating scan and over 18 years of age Able to provide informed consent (a translation service will be provided for women where English is not the first language);

Women recruited into Cohort B will have deferred consent taken to avoid interference with clinical care.

Exclusion Criteria:

* Pregnant woman under the age of 18 or wishing not to consent, withdrawing consent or lacking capacity.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Participants
Study Population: Pregnant women attending University Hospital of Wales Cardiff for their pregnancy care
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value of genomic sepsis-test biomarker in identifying participants with confirmed sepsis | 2 years
  New genomic sepsis-test biomarker tested to see if it compares to clinically known biomarkers in identifying sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ghazal, PHD, Principal Investigator — Cardiff University
Locations (1):
- Sir Geraint Evans, Cardiff University, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma S, Zaher S, Rodrigues PRS, Davies LC, Edkins S, Strang A, Chakraborty M, Watkins WJ, Andrews R, Parkinson E, Angelopoulos N, Moet L, Shepherd F, Davies KMM, White D, Oram S, Siddall K, Keeping V, Simpson K, Faggian F, Bray M, Bertorelli C, Bell S, Collis RE, McLaren JE, Labeta M, O'Donnell VB, Ghazal P. mSep: investigating physiological and immune-metabolic biomarkers in septic and healthy pregnant women to predict feto-maternal immune health - a prospective observational cohort study protocol. BMJ Open. 2022 Sep 17;12(9):e066382. doi: 10.1136/bmjopen-2022-066382. PMID 36115679